CLINICAL TRIAL: NCT04254640
Title: Efficacy and Safety of Cladribine in Combination With G-CSF,Low-dose Cytarabine and Aclarubicin in Newly Diagnosed Unfit Patients With Acute Myeloid Leukemia
Brief Title: Efficacy and Safety of Cladribine in Combination With CAG in Newly Diagnosed Unfit Patients With AML
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, wanghua, Director, Head of hematology, Principal Investigator, Clinical Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AML-2020
Record Dates: First submitted 2020-01-20; First posted 2020-02-05 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-01

CONDITIONS: Acute Myeloid Leukemia; Elderly Patients; Newly Diagnosed
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Cladribine; Aclarubicin; Granulocyte Colony-Stimulating Factor; Cytarabine

STUDY DESIGN:
Intervention Model Description: cladribine 5 mg/m2, d1-5; G-CSF 300 µg, d0-9; aclarubicin 10 mg, d3-6; cytarabine 10mg/ m2 q12h, SC, d3-9; 4 weeks per cycle.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- C-CAG (Experimental): cladribine 5 mg/m2, d1-5; G-CSF 300 µg, d0-9; aclarubicin 10 mg, d3-6; cytarabine 10mg/ m2 q12h, SC, d3-9; 4 weeks per cycle.
  Interventions: Drug: Cladribine Injection; Drug: Aclarubicin; Drug: G-CSF; Drug: cytarabine

INTERVENTIONS:
Drug: Cladribine Injection — Cladribine 5 mg/m2, intravenous drip,d1-5,4 weeks per cycle.
  Other Names: 2-chlorodeoxyadenosine
Drug: Aclarubicin — aclarubicin 10 mg, intravenous drip,d3-6,4 weeks per cycle.
  Other Names: aclarubicin hydrochloride
Drug: G-CSF — G-CSF 300 µg,subcutaneous injection, d0-9,4 weeks per cycle.
  Other Names: Granulocyte Colony-Stimulating Factor
Drug: cytarabine — cytarabine 10mg/ m2, subcutaneous injectionq,q12h, d3-9,4 weeks per cycle.
  Other Names: cytarabine hydrochloride

SUMMARY:
In this study, the investigators conducted a phase II trial that evaluated the efficacy and safety of cladribine in combination with modified CAG regimen (low-dose cytarabine and aclarubicin) in elderly patients with AML.

DETAILED DESCRIPTION:
The low-intensity chemotherapy were developed to reduce the early mortality and improve the benefit-risk ratio for longterm survival in elderly or unfit AML patients.Previous studies revealed that the standard dose of CAG regimen consisting of low-dose cytarabine and aclarubicin in combination with granulocyte colonystimulating factor (G-CSF) priming as an induction therapy was well-tolerated by patients and led to a complete remission (CR) rate of 50.0% in patients aged≥ 70 years. Cladribine (2-chlorodeoxyadenosine ) is a nucleoside analogue of anti-adenosine deaminase that has extensive antitumor activity in hematological tumor.The purine analog 2-CdA increases the uptake of Ara-C and the accumulation of its active cytotoxic metabolite 5α-triphosphate Ara-C (Ara-CTP) in leukemia cells. This finding suggests that synergy occurs between cladribine and cytarabine. In this study, the investigators conducted a phase II trial that evaluated the efficacy and safety of cladribine in combination with modified CAG regimen (low-dose cytarabine and aclarubicin) in unfit patients with AML.Patients will receive C-CAG regimen as follows: cladribine 5 mg/m2, d1-5; G-CSF 300 µg, d0-9; aclarubicin 10 mg, d3-6; cytarabine 10mg/ m2 q12h, SC, d3-9; 4 weeks per cycle. The participants are permitted to quit the study if complete remission (CR) was not achieved after two courses of chemotherapy.The participants will be treated for a total of six cycles unless disease progression or unacceptable side effects are observed or participants withdrew their consent.

ELIGIBILITY:
Inclusion Criteria:

Patients with:

1. a diagnosis of AML according to WHO 2016 classification (excluding acute promyelocytic leukemia) including secondary AML (after an antecedent hematological disease (e.g. MDS) and therapy-related AML
2. Patients 60 years and older.
3. Patients NOT eligible for standard chemotherapy, defined as hematopoietic cell transplantation comorbidity index (HCT-CI) ≥ 3 or Patients NOT eligible for standard chemotherapy for other reasons (wish of patient).
4. White blood cell (WBC) ≤ 10 x109/L (prior hydroxyurea allowed for a maximum of 5 days, stop 2 days before start cladribine treatment)
5. Adequate renal and hepatic functions unless clearly disease related as indicated by the following laboratory values:

   * Serum creatinine ≤ 221.7 µmol/L (≤ 2.5 mg/dL ), unless considered AML-related -Serum bilirubin ≤ 2.5 x upper limit of normal (ULN), unless considered AML-
   * related or due to Gilbert's syndrome
   * Alanine transaminase (ALT) ≤ 2.5 x ULN, unless considered AML-related
6. WHO performance status 0, 1 or 2.
7. Patient is willing and able to use adequate contraception during and until 5 months after the last protocol treatment.
8. Written informed consent.
9. Patient is capable of giving informed consent.

Exclusion Criteria:

1. Acute promyelocytic leukemia.
2. Acute leukemia's of ambiguous lineage according to WHO 2016
3. Patient has symptomatic central nervous system (CNS) leukemia (NO routinely lumbar puncture required to investigate CNS involvement)
4. Blast crisis of chronic myeloid leukemia.
5. Diagnosis of any previous or concomitant malignancy is an exclusion criterion:
6. except when the patient completed successfully treatment (chemotherapy and/or surgery and/or radiotherapy) with curative intent for this malignancy at least 6 months prior to randomization. OR
7. except for basal and squamous cell carcinoma of the skin or in situ carcinoma of the cervix
8. Patients previously treated for AML (any antileukemic therapy including investigational agents), a short treatment period ( ≤ 5 days) with Hydroxyurea is allowed
9. Current concomitant chemotherapy, radiation therapy, or immunotherapy; other than hydroxyurea
10. Concurrent severe and/or uncontrolled medical condition (e.g. uncontrolled diabetes, infection, hypertension, pulmonary disease etc.)
11. Cardiac dysfunction as defined by:

    * Myocardial infarction within the last 3 months of study entry, or
    * Reduced left ventricular function with an ejection fraction < 40% as measured by MUGA scan or echocardiogram or
    * Unstable angina or
    * New York Heart Association grade IV congestive heart failure or
    * Unstable cardiac arrhythmias.
12. History of stroke or intracranial hemorrhage within 6 months prior to randomization.
13. Patient has a history of human immunodeficiency virus or active infection with Hepatitis C or B.
14. Patients known to be pregnant
15. Patients with a history of non-compliance to medical regimens or who are considered unreliable with respect to compliance.
16. Patients with any serious concomitant medical condition which could, in the opinion of the investigator, compromise participation in the study.
17. Patients who have senile dementia, mental impairment or any other psychiatric disorder that prohibits the patient from understanding and giving informed consent.
18. Any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2021-03-01 (Estimated); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Cumulative Complete Remission (CR) / CR with incomplete blood count (CRi) rate | At the end of Cycle 2 (each cycle is 28 days)
  Cumulative CR/CRi rate during 2 cycles

SECONDARY OUTCOMES:
Safety and tolerability of Cladribine in Combination With CAG determined by the type, frequency, severity and relationship of adverse events to study treatment | 1 years
  Safety and tolerability of Cladribine in Combination With treatment for CAG for AML (type, frequency, severity and relationship of adverse events to study treatment).
Event free survival (EFS) | 5 years
  The time from registration to induction failure, death or relapse whichever occurs first
Overall survival (OS) | 5 years
  The time from the date of registration to the date of death, whatever the cause. Patients still alive at the date last contact will be censored.
Prognostic value of MRD | 9 months and at relapse
  Assessment of the prognostic value of Minimal Residual Disease (MRD) by flowcytometry or PCR

CONTACTS AND LOCATIONS:
Overall Officials: wang hua, MD., Principal Investigator — sun yat-sun university cancer
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China